CLINICAL TRIAL: NCT05917600
Title: Impact of Advanced Practical Nursing Intervention Versus Usual Care on Hypertension Control: Study Protocol for an Open-label Randomized Controlled Trial
Brief Title: Impact of Advanced Practical Nursing Intervention Versus Usual Care on Hypertension Control
Acronym: iIPA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: APHP230450; 2023-A00189-36 (Other: ANSM)
Record Dates: First submitted 2023-06-14; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-05

CONDITIONS: Hypertension
Keywords: Advanced practice nurse; Hypertension; Therapeutic adherence; Trial
MeSH Terms: conditions — Hypertension; Treatment Adherence and Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): The interventional group meets an Advanced Practice Nurses (APN) between the ambulatory hospitalization (AH) and the MD consultation
  Interventions: Other: APN intervention
- Control group (No Intervention): The control group of patients keeps a traditional follow-up (ambulatory hospitalization (AH) then consultation with a MD)

INTERVENTIONS:
Other: APN intervention — Advanced Practice Nurses (APN) intervention between the ambulatory hospitalization (AH) and the MD consultation
  APN intervention is divided into five main steps:
  * clinical and paraclinical examinations,
  * appraisal of patient's knowledge,
  * health education on hypertension and treatments,
  * setting a written medication plan with the patient to invest him in his management with adjusting or renewing treatments identically if necessary
  * decision-making balance between the benefits and risks of non-adherence to medication. A time is scheduled at the end of the intervention to let the patient ask questions or express his difficulties if he needs to.
  Arms: Interventional group

SUMMARY:
Hypertension is the most frequent chronic pathology in France and in the world. It is one of the main modifiable cardiovascular risk factors. In France, 50% of treated hypertensives are uncontrolled and only 30% of treated patients are fully adherent to their antihypertensive treatment. Poor adherence to drug treatments is considered as one of the main causes of non-control of hypertension.

Since 2018, a new profession has entered the French healthcare system: Advanced Practice Nurses (APN). They have many broad skills, at the interface of nursing and medical exercises.

The purpose of this interventional study is to assess the impact of APN on blood pressure (BP) control in the context of usual care of hypertension thanks to a better adhesion of patients and a better therapeutic alliance.

The hypothesis formulated is that an individual APN intervention, included in a usual hypertension management, improves BP control.

DETAILED DESCRIPTION:
This study will be a prospective, open-label, randomized 1-to-1 and monocentric trial, conducted at the Diagnosis and Therapeutic Center of the Hôtel-Dieu University Hospital, Assistance Publique - Hôpitaux de Paris, France.

Recruitment will be conducted during the ambulatory hospitalization. After the signature of the consent form, the randomization will be conducted during the ambulatory hospitalization. All recruited patients will be randomized.

According to the randomization, the odd-numbered participants will constitute the "usual care" group, and the even-numbered patients will constitute the "intervention" group.

The "usual care" group will keep a traditional follow-up: ambulatory hospitalization then consultation with a MD within approximately 2 to 12 months.

The "intervention" group will meet the APN between the ambulatory hospitalization and the MD consultation, within 1 to 6 months.

The participants will get their study appointment(s) (MD consultation +/- APN intervention) at the end of the ambulatory hospitalization according to their allocation.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age,
* Essential Hypertension
* Hypertension management in Hôtel-Dieu Hospital
* Ability to provide a written informed consent.

Exclusion Criteria:

* Have already benefited from an APN follow-up before the day of inclusion
* Being under guardianship or curatorship
* Pregnant patient
* Beneficiary of the AME (state medical aid)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Blood pressure control | Medical consultation, from 2 months to 12 months after inclusion
  Blood pressure < 140/90 mmHg

SECONDARY OUTCOMES:
Rate of patients who brought HBPM to consultation | Medical consultation, from 2 months to 12 months after inclusion
  Ability to realize a home blood pressure measurement Blood pressure control in home blood pressure measurement (HBPM)
Number of measurements | Medical consultation, from 2 months to 12 months after inclusion
  Ability of HBPM Quality of the HBPM : Number of measurements carried out over 3 days (18 measurements over 3 days according to protocol) then divided into 4 categories: performance (18 measurements), average performance (17 to 15 measurements), average performance (14 to 12 measurements or less), poor performance (11 measures or less).
Rate of Blood pressure control | Medical consultation, from 2 months to 12 months after inclusion
  Difference between inclusion and the Medical consultation, from 2 months to 12 months after inclusion
Rate of therapeutic adjustments | Medical consultation, from 2 months to 12 months after inclusion
  Rate of therapeutic adjustments due to side effects
Rate of therapeutic adjustments | Medical consultation, from 2 months to 12 months after inclusion
  Rate of therapeutic adjustments due to uncontrolled hypertension
Rate of therapeutic adjustments | Medical consultation, from 2 months to 12 months after inclusion
  Rate of therapeutic adjustments : other reason

CONTACTS AND LOCATIONS:
Overall Officials: Jacques BLACHER, MD, PhD, Principal Investigator — Diagnosis and Therapeutic Center, Hôtel-Dieu Hospital, Assistance Publique-Hôpitaux de Paris; Juliette VAY-DEMOUY, MSc, PhD, Study Director — Diagnosis and Therapeutic Center, Hôtel-Dieu Hospital, Assistance Publique-Hôpitaux de Paris
Locations (1):
- Diagnosis and Therapeutic Center, Hôtel-Dieu Hospital, Paris, IDF, France

IPD SHARING:
Plan to Share IPD: Undecided